CLINICAL TRIAL: NCT07106684
Title: A Prospective, Single-Arm, Phase II Study of Autologous Stem Cell Transplantation Combined With BCMA CAR-T Therapy Followed by GPRC5D/CD3 Bispecific Antibody Maintenance in Transplant-Eligible Patients With Primary Plasma Cell Leukemia
Brief Title: ASCT Combined With BCMA CAR-T and GPRC5D/CD3 BiTEs Maintenance for Transplant-Eligible Primary Plasma Cell Leukemia
Acronym: CAREMM-004
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2025048
Record Dates: First submitted 2025-07-30; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Multiple Myeloma, Plasma Cell Leukemia
Keywords: Plasma cell leukemia; CAR-T; ASCT; BiTEs
MeSH Terms: conditions — Multiple Myeloma; Leukemia, Plasma Cell; Bites and Stings

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ASCT Combined With BCMA CAR-T and GPRC5D/CD3 BiTEs Maintenance (Experimental): Patients will receive induction therapy, undergo ASCT followed by BCMA CAR-T infusion. Three month after CAR-T cell infusion, patients will begin GPRC5D/CD3 BiTEs maintenance therapy for ≥2 years.
  Interventions: Procedure: Autologous hematopoietic stem cell transplantation; Biological: BCMA CAR-T; Drug: GPRC5D/CD3 BiTEs

INTERVENTIONS:
Procedure: Autologous hematopoietic stem cell transplantation — Patients receive transplantation conditioning followed by autologous hematopoietic stem cell transplantation after successful stem cell mobilization and collection.
Biological: BCMA CAR-T — Patients will receive BCMA CAR-T single dose (3.0 x 10^6 cells /kg) infusion 3 days after ASCT.
Drug: GPRC5D/CD3 BiTEs — Patients will receive GPRC5D/CD3 BiTEs maintenance therapy at a dose of 54 μg/kg every 4 weeks, starting 3 months after BCMA CAR-T infusion and continuing for at least 2 years

SUMMARY:
This is a prospective, single-arm, phase II study to evaluate the efficacy and safety of autologous stem cell transplantation combined with BCMA CAR-T therapy followed by GPRC5D/CD3 bispecific antibody maintenance in transplant-eligible patients with primary plasma cell leukemia.

DETAILED DESCRIPTION:
All subjects will receive standard induction therapy for up to four cycles prior to screening. Following response evaluation, those who meet the inclusion criteria will be enrolled. Enrolled patients will undergo autologous stem cell transplantation (ASCT) combined with BCMA CAR-T cell therapy, followed by GPRC5D/CD3 bispecific antibody therapy.

Patients who achieve a stringent complete response (sCR) and sustained MRD negativity (≥12 months) will receive maintenance therapy for 24 months, and may then enter a treatment-free observation phase. Patients who experience MRD resurgence or loss of response during observation will resume maintenance therapy.

Patients who do not achieve both sCR and sustained MRD negativity (≥12 months) will continue GPRC5D/CD3 bispecific antibody therapy until disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years and ≤ 70 years.
2. Participants with documented newly-diagnosed primary plasma cell leukemia according to IMWG diagnostic criteria.
3. Measurable disease at screening, defined as: Serum M-protein level ≥1.0 g/dL or urine M-protein level ≥200 mg/24 hours; or Light chain MM without measurable disease in serum or urine: serum Ig free-light chain (FLC) ≥10 mg/dL and abnormal serum Ig kappa lambda FLC ratio.
4. Patients deemed eligible for high-dose chemotherapy with ASCT.
5. Tumor cells were BCMA and GPRC5D positive.
6. Serum total bilirubin <2 x upper limit of normal (ULN), serum AST and ALT <3 x ULN, creatinine clearance ≥ 30mL/min (Cockroft-Gault formula).
7. Informed Consent/Assent: All subjects have the ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

1. Active amyloidosis.
2. Central nervous system involvement.
3. Prior BCMA-targeted therapy or CAR-T therapy.
4. Active hepatitis B or hepatitis C virus infection.
5. Known HIV infection.
6. Life expectancy <6 months.
7. Woman who are pregnant or breastfeeding
8. Evidence of uncontrolled dysfunction of heart, lung, brain, and other important organs.
9. Any other conditions that are not eligible for the trial in the judgement of the principal investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-08-10 (Estimated); Primary Completion 2027-08-01 (Estimated); Study Completion 2029-08-01 (Estimated)

PRIMARY OUTCOMES:
Sustained MRD-negative rate | Up to 2 year
  Rate of patients achieving sustained MRD negativity for more than 12 months
MRD negativity rate | Up to 2 years
  Rate of patients achieving MRD negativity

SECONDARY OUTCOMES:
Safety and Tolerability | Up to 2 year
  The incidence of treatment-emergent adverse events (TEAEs)
Complete response rate (CRR) | Up to 2 years
  CR or better is defined as percentage of participants who achieve a CR response or Stringent Complete Response (sCR) response accoording to the IMWG criteria
Progression free survival (PFS) | Up to 3 year
  Progression free survival is defined as the time from the date of diagnosis to the date of first documented PD, as defined in the IMWG criteria, or death due to any cause, whichever occurs first
Overall survival (OS) | Up to 5 year
  Overall survival is defined as the time from the date of diagnosis to the date of death due to any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Hematology and Blood Diseases Hospital Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No